CLINICAL TRIAL: NCT03474146
Title: "Comparative Evaluation of Antiplaque and Antigingivitis Efficacy of Ocimum Sanctum (Tulsi) Extract Mouthrinse With 0.12% Chlorhexidine Mouthrinse - an in Vitro and in Vivo Study."
Brief Title: Comparative Evaluation of Antiplaque and Antigingivitis Efficacy of Ocimum Sanctum (Tulsi) Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Dr. Pratik kumar Ashok bhai Chaudhari, Postgraduate student, Government College of Dentistry, Indore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 32/IEC/SS/2017
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Periodontal Diseases; Gingivitis; Periodontitis
Keywords: Mouthrinse; Ocimum sanctum; Periodontal Diseases; Tulsi
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Periodontitis | interventions — holy basil leaf extract; chlorhexidine gluconate; Chlorhexidine; Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ocimum sanctum extract as mouthrinse (Experimental): 10ml mouthrinse was rinsed for 60sec twice a daily for 03 weeks.
  Interventions: Other: Ocimum sanctum
- Chlorhexidine Gluconate as mouthrinse (Active Comparator): 10ml mouthrinse was rinsed for 60sec twice a daily for 03 weeks.
  Interventions: Other: Chlorhexidine Gluconate
- Propylene Glycol as mouthrinse (Placebo Comparator): 10ml mouthrinse was rinsed for 60sec twice a daily for 03 weeks.
  Interventions: Other: Propylene Glycol

INTERVENTIONS:
Other: Ocimum sanctum — Ocimum sanctum (known as Tulsi, Holy basil) is natural herb which is known for its broad spectrum medicinal properties. Ocimum sanctum is one of the best examples of Ayurveda's holistic lifestyle approach to health. It is also been well practiced in traditional medicine in India and south Asian region. Literature showed that Ocimum sanctum extract have significant anti-gingivitis and anti-inflammatory effect as mouthrinse.
  Other Names: Tulsi; Holy Basil
  Arms: Ocimum sanctum extract as mouthrinse
Other: Chlorhexidine Gluconate — Chlorhexidine Gluconate (C34H54Cl2N10O14) is a bisbiguanide formulation with cationic properties. Chlorhexidine over a period of over 40 years has been thoroughly investigated and successfully used as plaque control agent in dental practice. A literature review, highlighting chlorhexidine as not only a plaque control agent but also as an effective antimicrobial agent and its wider application in variety of oral disorders in various formulations.
  Other Names: Chlorhexidine
  Arms: Chlorhexidine Gluconate as mouthrinse
Other: Propylene Glycol — Propylene glycol or 1,2-dihydroxypropane or 1,2-propanediol, is a clear, colourless, viscous, practically odourless liquid with a density of 1.038 g/cm³ at 20 °C and a molecular weight of 76.095. It is miscible with water, acetone and chloroform. It is miscible in water. Propylene glycol is commonly used as an excipient in a variety of drugs and it is also authorised in food products and cosmetics.
  Arms: Propylene Glycol as mouthrinse

SUMMARY:
Chlorhexidine is considered as gold standard for its antiplaque and antigingivitis efficacy till date but it has got many side effects. So it is need of the hour that investigators will find some substitute having similar antiplque and antigingivitis efficay but have less or no adverse effects. so in this study investigators planned to do "Comparative evaluation of antiplaque and antigingivitis efficacy of ocimum sanctum (tulsi) extract mouthrinse with 0.12% chlorhexidine mouthrinse.

DETAILED DESCRIPTION:
Title:

"Comparative evaluation of antiplaque and antigingivitis efficacy of ocimum sanctum (tulsi) extract mouthrinse with 0.12% chlorhexidine mouthrinse - an in vitro and in vivo study."

Aims And Objectives:

1. To evaluate the antimicrobial activity of Ocimum sanctum (Tulsi) extract by Sensitivity testing, Minimum Inhibitory Concentration, Minimum Bactericidal Concentration, and Time kill curve -In Vitro study.
2. To evaluate the Antiplaque and Antigingivitis effect of the Ocimum sanctum (Tulsi) by recording Modified Gingival Index and Modified Plaque Index in patients with Chronic Generalized Gingivitis and Mild Chronic Generalized Periodontitis -In Vivo study.
3. Clinical evaluation and comparison of the Antiplaque and Antigingivitis effect of the Ocimum sanctum (Tulsi) with 0.12% Chlorhexidine and vehicle.
4. To see the topical beneficial and/or harmful side effects of Ocimum sanctum extract, if any.

Study Design:

Prospective randomized controlled Trial- Randomized Comparative Study

Methodology (Material & Methods):

The present study will have following parts:

1. Procurement of extract and formulation of mouthrinse: Ocimum sanctum (Tulsi) extract has been purchased from the ISO (International Organization for Standardization) Certified shop. The desired mouthrinse will be formulated under the guidance of Department of Pharmacology, Mahatma Gandhi Memorial Medical College, Indore (M.P.)
2. In vitro study: Sensitivity testing, Minimum Inhibitory Concentration (MIC) and Minimum Bactericidal Concentration (MBC), of Ocimum sanctum will be determined against following microorganisms: Porphyromonas gingivalis, Prevotella intermedia, Fusobacterium nucleatum, Aggregatibacter actinomycetemcomitans, Capnocytophaga, Tannerella forsythia, Pseudomonas aeruginosa, and other microorganisms.
3. In vivo study: This study has been planned and would be conducted in the Department of Periodontology, Govt. College of Dentistry, Indore, Madhya pradesh, India. In this study, participants with Chronic Generalized Gingivitis and Mild Chronic Generalized Periodontitis would be randomly selected from outdoor patients. A minimum 90 Recruited participants will be divided into three equal groups randomly. (Parallel design, case control, Randomized Comparative Study).

Group A: (Test group) (n=30) Ocimum sanctum extract as mouthrinse. Group B: (Positive control group) (n=30) 0.12% Chlorhexidine as mouthrinse. Group C: (control group) (n=30) Vehicle as the mouthrinse. All the three solutions would be prepared under the valuable guidance of Department of Pharmacology, Mahatma Gandhi Memorial Medical College, Indore (M.P.) and will be kept in coded containers. All the participants in each group would be advised to use their respective mouth rinses twice daily with proper swishing action for a minute, after brushing their teeth (in the morning and before going to bed). To maintain standardization, similar toothbrushes and dentifrices will be provided to all the participants (free of cost) and standard tooth brushing techniques will be demonstrated.

Written consent will be obtained from each participants, and then followed by case history taking along with clinical examination by recording various periodontal parameters taken in the study.

Following clinical periodontal parameters are to be recorded at baseline, at 1 week, at 2 weeks, and at 3 weeks:

1. Modified Gingival Index
2. Modified Plaque Index

Sample Size:

Minimum 90 patients with Generalized Chronic Gingivitis or Mild Generalized Chronic Periodontitis will be selected. Participants will be divided into 03 different groups, n=30 participants in each group by computer generated table of random numbers.

Data Collection And Methods:

Cases with Generalized Chronic Gingivitis or Mild Generalized Chronic Periodontitis of either sex and the age group 18-40 years who abide by approved protocol guidelines and are ready to give written informed consent will be selected randomly from OPD (outpatient department) of The Department of Periodontology, Govt. College of Dentistry, Indore (M.P.). The selected participants will be equally divided into three groups, by computer generated random number table.

ELIGIBILITY:
Inclusion criteria

* Cases with generalized chronic gingivitis or cases with mild generalized chronic periodontitis patients of any sex.
* Systemically healthy individuals.
* Participants having >20 teeth.
* Participants in the age group of 18-40 years, who abide by approved protocol guidelines, and are ready to give written informed consent.

Exclusion criteria

* Any known systemic disease which has effects on periodontium such as diabetes, cardiovascular, cancer etc.
* Participants on anti-inflammatory, perioceutics, antibiotics, steroids, cytotoxic and drugs since 03 months.
* Participants who have known allergy to material used for the study.
* Pregnant and lactating mothers.
* Participants had undergone any kind of nonsurgical and/or surgical periodontal therapy earlier, in past 6 months.
* Tobacco users (smoke and smokeless) and alcoholics.
* Participants wearing any form of intraoral prosthesis or appliance.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Modified Gingival Index | Change from baseline Gingival index at 03 weeks
  The Modified Gingival Index (Lobene, Weatherford, Ross, Lamm, 1986) was recorded based on following criteria: 0 - Absence of inflammation. 1 - Mild inflammation or with slight changes in color and texture but, not in all portions of marginal or papillary gingiva. 2 - Mild inflammation, such as the preceding criteria, in all portions of marginal or papillary gingiva. 3 - Moderate, bright surface inflammation, erythema, edema, and/or hypertrophy of marginal or papillary gingiva. 4 - Severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration. Modified Gingival Index = Total score of all teeth / no. of sites

SECONDARY OUTCOMES:
Modified Plaque Index | Change from baseline Plaque index at 03 weeks
  Plaque Index (Turesky, Gilmore, Glickman modification of Quigely Hein Index, 1970) Scoring was as follows: 0 - No plaque/debris. 1 - Separate flecks of plaque at the cervical margin of the tooth. 2 - A thin continuous band of plaque (up to 1mm) at the cervical margin of the tooth. 3 - A band of plaque wider than 1 mm but covering less than one third of the crown of the tooth. 4 - plaque covering at least one third but less than two thirds of the crown of the tooth. 5 - Plaque covering two third or more of the crown of the tooth. Plaque Index = Total score / no. of surfaces examined

OTHER OUTCOMES:
Minimum Inhibitory Concentration (MIC) | Up to 24 hours
  Minimum inhibitory concentration (MIC) is the lowest concentration of a chemical which prevents visible growth of a bacterium. Tested against following periopathogens: Porphyromona sgingivalis, Prevotella intermedia, fusobacteriumnucleatum, Aggregatibacter actinomycetemcomitans, Capnocytophaga, Tanerella forsythia, Pseudomonas aeruginosa, Streptococcus mutans, E. fecalis, and Candida.
Minimum bactericidal concentration (MBC) | Up to 24 hours
  Minimum bactericidal concentration (MBC) is the concentration resulting in microbial death as defined by the inability to re-culture bacteria. Tested against following periopathogens: Porphyromona sgingivalis, Prevotella intermedia, fusobacteriumnucleatum, Aggregatibacter actinomycetemcomitans, Capnocytophaga, Tanerella forsythia, Pseudomonas aeruginosa, Streptococcus mutans, E. fecalis, and Candida.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Subhash Garg, M.D.S., Study Director — Govt. College of Dentistry, Indore, Madhya pradesh, India
Locations (1):
- GCD Indore, Indore, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta D, Bhaskar DJ, Gupta RK, Karim B, Jain A, Singh R, Karim W. A randomized controlled clinical trial of Ocimum sanctum and chlorhexidine mouthwash on dental plaque and gingival inflammation. J Ayurveda Integr Med. 2014 Apr;5(2):109-16. doi: 10.4103/0975-9476.131727. PMID 24948862
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376